CLINICAL TRIAL: NCT07226167
Title: Evaluating the Impact of Hearing Aid Signal Enhancement Algorithms in Real-World Contexts
Brief Title: Hearing Aid Benefit in Real-World Noisy Environments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-1586; FA (Other: UW Madison); UWMSN | L&S | Communication Sc (Other: UW Madison); Protocol Version 11/25/25 (Other: UW Madison)
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Hearing Aid; Hearing Loss, Bilateral Sensorineural; Hearing Loss, Adult-Onset
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hearing aid + smartphone surveys (Experimental): Participants will use study-provided hearing aids
  Interventions: Device: Hearing aid

INTERVENTIONS:
Device: Hearing aid — Participants will use study-provided hearing aids for 15 minutes, 7-10 times for a week.

SUMMARY:
Researchers are doing this study to understand why hearing aids often work well in controlled laboratory settings but don't provide the same level of benefit in everyday noisy environments. The questions they hope to answer are:

* What factors contribute to hearing aid benefit in noisy environments
* What factors limit hearing aid benefit
* How do real-world factors interact with common hearing aid settings

Participants will complete:

* Hearing and listening tests
* Memory and attention assessment
* Surveys on their Smartphone

DETAILED DESCRIPTION:
This is study investigates how hearing aid signal processing algorithms and environmental factors in listening situations interact to affect listening outcomes. A crossover design is used to assess speech perception, listening effort, and user satisfaction across diverse acoustic contexts.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Symmetrical, bilateral, adult onset, sensorineural hearing loss
* Experienced hearing aid users (> 3 months)

Exclusion Criteria:

* Under 18 years old
* Conductive or mixed hearing loss
* Asymmetrical or unilateral hearing loss
* Pre-lingual or childhood hearing loss onset
* No hearing aid experience

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Compare effectiveness of hearing aid signal enhancement on speech perception | 1 week
  Participants will hear 3 different, 5 minute listening scenarios and answer the same survey questions for each. They will rate perception from 0% (understood nothing) to 100% (understood everything). Percentages will be compared across the 3 scenarios.
Compare effectiveness of hearing aid signal enhancement on listening effort | 1 week
  Participants will hear 3 different, 5 minute listening scenarios and answer the same survey questions for each. They will rate how hard they had to work to understand what was said from 0% (no effort) to 100% (extremely hard). Percentages will be compared across the 3 scenarios.
Compare effectiveness of hearing aid signal enhancement on listening comfort | 1 week
  Participants will hear 3 different, 5 minute listening scenarios and answer the same survey questions for each. They will rate how comfortable it was to listen from 0% (very comfortable) to 100% (very uncomfortable). Percentages will be compared across the 3 scenarios.
Compare effectiveness of hearing aid signal enhancement on sound quality | 1 week
  Participants will hear 3 different, 5 minute listening scenarios and answer the same survey questions for each. They will rate the sound quality from 0% (very poor) to 100% (excellent). Percentages will be compared across the 3 scenarios.
Compare effectiveness of hearing aid signal enhancement on sound location | 1 week
  Participants will hear 3 different, 5 minute listening scenarios and answer the same survey questions for each. They will rate how easy it was to tell where the sound was coming from, from 0% (could not tell) to 100% (very easy). Percentages will be compared across the 3 scenarios.
Compare effectiveness of hearing aid algorithms based on location | 1 week
  Participants will complete the same survey questions for all three algorithms. Participants will select which option best describes the environment they are in when completing the hearing survey.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Jorgensen, AuD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes